CLINICAL TRIAL: NCT03800069
Title: Biomedical Device Trial of Validation of Point of Care Liver Function Tests
Brief Title: Validation of Point of Care Liver Function Tests
Status: Terminated | Type: Observational
Why Stopped: scheduling complexities
Sponsor: University of Pennsylvania (Other)
Collaborators: Group K Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 829476
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Liver Diseases; Healthy; Cirrhosis, Liver; Fibrosis
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: A finger stick sample is collected and tested on the study device.
  Interventions: Device: Group K Diagnostic point of care device

INTERVENTIONS:
Device: Group K Diagnostic point of care device — Arm 1 will have a finger prick sample collected to test the ability of Group K Diagnostic point of care device and app to identify liver function values.

SUMMARY:
This study is testing the accuracy of a point of care device that tests liver function within 20 minutes. The target population will be any adult who had liver function tests ordered and to be drawn on the same day as enrollment.

DETAILED DESCRIPTION:
Outpatient diagnostics are slow and expensive due to turnaround times, complex workflows and high cost. Sometimes patients do not make it to laboratory testing if a lab is not available on site. Delays in testing can affect medical outcomes or patients can be lost to follow up.

Group K developed a paper microfluidic platform with an accompanying mobile application(app). The paper microfluidic device is a simple, inexpensive wax backed device with three testing areas. These areas have a mix of dried proprietary reagents that when combined with a patients drop of blood, or in the future, saliva or urine, will produce results in a color change. An app is then used to interpret the color change and output results to a doctor. The target population is adults who have an indication to collect a liver function panel that will be drawn on the same day as their clinic visit or during their inpatient hospital

ELIGIBILITY:
Inclusion Criteria:

* Have a liver function testing for the required 6 tests completed (Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), albumin, bilirubin, and total protein)
* 18 years or older

Exclusion Criteria:

* Inadequate blood sample obtained from finger stick
* Inconclusive liver function testing
* Not all 6 liver tests completed on the same sample
* Liver tests not drawn for normal method at same time as finger stick.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from inpatient and clinic setting at The Hospital of the University of Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Regression curve and correlation coefficient | 1 year
  Each data point will represent one observation or one test run. The investigators will use regression methods to determine the linear relationship between standard lab results and Group K diagnostic's device.

SECONDARY OUTCOMES:
The consistent accuracy of the diagnostic device | 1 year
  Lowest level frequency of detection must be detected 90% of the time. This will become the functional lower limit. The same with the highest level of frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Khungar, MD, MSc, Principal Investigator — Director of Inpatient Hepatology
Locations (1):
- The Hospital of the University of Pennslyvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03800069/Prot_000.pdf
  • Informed Consent Form (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03800069/ICF_001.pdf